CLINICAL TRIAL: NCT02850068
Title: Geniculate Artery Embolization for the Treatment of Knee Pain Secondary to Osteoarthritis
Brief Title: Geniculate Artery Embolization for the Treatment of Knee Pain
Acronym: GAE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-1969
Record Dates: First submitted 2016-07-27; First posted 2016-07-29 (Estimated); Results first posted 2019-08-20 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-04

CONDITIONS: Osteoarthritis Of Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Geniculate Artery Embolization (Experimental): Patients in this study will receive the geniculate artery embolization (GAE) procedure. The primary aims will be to determine if geniculate artery embolization (GAE) will reduce pain and disability (resulting from pain, stiffness and difficulty performing daily activities) caused by knee osteoarthritis (OA).
  Interventions: Device: Geniculate Artery Embolization

INTERVENTIONS:
Device: Geniculate Artery Embolization — Geniculate artery embolization (GAE) is a new procedure that is being used to reduce pain and disability (resulting from pain, stiffness and difficulty performing daily activities) caused by knee osteoarthritis (OA). Embolization is a procedure where physicians intentionally block the blood vessels to specific areas of the body to prevent blood flow to that region. By doing this, the decrease in blood flow will decrease the size of the area of interest. In this case, the goal is to decrease the size of inflammatory tissue around the knee, resulting in improvement of pain, stiffness and difficulty performing daily activities from OA.
  Other Names: Embozene Microspheres

SUMMARY:
This study is to test a new treatment method, geniculate artery embolization (GAE), to reduce the severity of pain and disability caused by knee osteoarthritis.

DETAILED DESCRIPTION:
Purpose: The primary aims of this study are to determine if geniculate artery embolization (GAE) will reduce the severity of pain as well as global disability (resulting from the combination of pain, stiffness and difficulty performing daily activities) caused by knee OA and if it can be performed safely. The secondary aim is to determine if GAE can result in the decreased necessity for ongoing conservative OA therapies such as medication therapy and joint injections.

Participants: Twenty patients with knee osteoarthritis resulting in knee pain that is refractory to conservative therapies, who are not planning to undergo surgery within 6 months.

Procedures (methods): This will be an open label 24-month pilot study with a small population undergoing GAE to determine safety and efficacy. Clinical procedures and evaluations will consist of a preoperative screening assessment to determine if the potential study subject meets the inclusion and exclusion criteria, enrollment, surgical procedure for geniculate artery embolization, and follow-up visits at 24 hours, 1, 3 & 6 months. An MRI will be performed at the 1-month visit to detect a change in synovial vascularity and to exclude complication.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe knee pain (visual analog scale (VAS) > 50 mm), and
* Pain refractory to at least 3 months* of conservative therapies (anti-inflammatory drugs, or physical therapy, or muscle strengthening, or intra-articular injections), and
* Kellgren-Lawrence grade 1, 2 or 3 on radiograph of the knee.

Exclusion Criteria:

* Current local infection, or
* Life expectancy less than 6 months, or
* Known advanced atherosclerosis, or
* Rheumatoid or infectious arthritis, or
* Prior knee surgery, or
* Uncorrectable coagulopathy including international normalized ratio (INR) > 2.5 or platelets < 30,000, or
* Iodine allergy resulting in anaphylaxis, or
* Renal dysfunction as defined by serum creatinine >1.6 dl/mg obtained within the past 30 days.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-01-25 (Actual); Primary Completion 2018-08-03 (Actual); Study Completion 2018-08-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ari Isaacson, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (2):
- United States (2):
  - UNC Hospitals, Chapel Hill, North Carolina
  - Vascular Institute of Virginia, Woodbridge, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Geniculate Artery Embolization
Started | 20
Completed | 0
Not Completed | 20

BASELINE CHARACTERISTICS:
Arm/Group | Geniculate Artery Embolization
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 20
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Patient Function (Units on a Scale)
Description: Western Ontario and McMaster University Osteoarthritis Index will be used to measure function. This is a score derived from a questionnaire in which the patient answers questions regarding rheumatic symptoms, stiffness, pain and how it affects the ability to function. Participants are asked to rate each question on a scale from 0 to 4 (0 = None, 1 = Slight, 2 = Moderate, 3 = Very, 4 = Extremely) for the level of difficulty to complete each task. The categories are then totaled for an overall score out of 96. Higher values indicate greater levels of pain, stiffness, and functional limitations.
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Geniculate Artery Embolization
Number analyzed (Participants) | 20
units on a scale | 31 [18 to 44]

2. Primary Outcome: Patient Pain (mm)
Description: The pain intensity is assessed using a visual analogue scale (VAS), which is a horizontal line 100 mm in length. Subjects mark the VAS with a single vertical line to indicate their current pain level, with 0 mm representing "No Pain" and 100 mm representing "Worst Possible Pain".
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: mm
Arm/Group | Geniculate Artery Embolization
Number analyzed (Participants) | 20
mm | 31 [17 to 45]

3. Secondary Outcome: Reduction in Medication (Percentage of Participants With a Reduction in Medication Therapy at Month 6)
Description: Reduction in the number or strength of previously initiated OA medical therapy (e.g. NSAIDs) at 6 months follow-up, which will be summarized using counts and simple statistics (percentage of participants with a reduction in medication therapy at month 6 months).
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Geniculate Artery Embolization
Number analyzed (Participants) | 20
percentage of participants | 65 [41 to 85]

4. Other Pre Specified Outcome: Patient Complications (Number of Participants With Complications at Month 6)
Description: The number and description of complications, adverse events, or poor outcomes that are secondary to the GAE procedure, which will be summarized using counts and simple statistics (number of participants with complications at month 6)
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Geniculate Artery Embolization
Number analyzed (Participants) | 20
Participants | 16

ADVERSE EVENTS:
Time Frame: 6 months following procedure
Arm/Group | Geniculate Artery Embolization
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 16/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Geniculate Artery Embolization (N=20)
small access site hematoma (Skin and subcutaneous tissue disorders) | 1 (1) — Small hematoma at site of access for procedure
skin discoloration without ulcer that resolved by 3-months follow-up evaluation without intervention (Skin and subcutaneous tissue disorders) | 13 (13)
great toe plantar numbness that resolved within 2 weeks (Nervous system disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2017-09-08): https://cdn.clinicaltrials.gov/large-docs/68/NCT02850068/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2017-05-31): https://cdn.clinicaltrials.gov/large-docs/68/NCT02850068/Prot_SAP_001.pdf